CLINICAL TRIAL: NCT04101370
Title: Two-way Crossover, Open-label, Single-dose, Bioequivalence Study of Bosentan (LLC "GEROPHARM", Russia) 125 mg Tablets Immediate Release (IR )Versus Tracleer® (Actelion Pharmaceuticals Ltd., Switzerland) 125 mg Tablets IR in Normal Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Bosentan 125 mg Tablets Immediate Release (IR) Versus Tracleer® 125 mg Tablets IR In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BOZ-501
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-03

CONDITIONS: Bioequivalence
Keywords: AUC; Cmax; Pharmacokinetics; bosentan; fasting
MeSH Terms: conditions — Fasting | interventions — Bosentan; Tablets

STUDY DESIGN:
Intervention Model Description: Crossover Assignment two-way crossover
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bosentan (Experimental): Single administered dose of Bosentan (125 mg tablet immediate release) in a fasting condition
  Interventions: Drug: Bosentan 125 mg
- Tracleer® (Active Comparator): Single administered dose of Tracleer® (125 mg tablet immediate release) in a fasting condition
  Interventions: Drug: Tracleer 125Mg Tablet

INTERVENTIONS:
Drug: Bosentan 125 mg — Single administered dose of Bosentan (125 mg tablet immediate release) in a fasting condition
  Other Names: bosentan
  Arms: Bosentan
Drug: Tracleer 125Mg Tablet — Single administered dose of Tracleer® (125 mg tablet immediate release) in a fasting condition
  Other Names: bosentan
  Arms: Tracleer®

SUMMARY:
Bioequivalence Study of 2 formulation of bosentan (Bosentan GEROPHARM vers. Tracleer® Actelion)

DETAILED DESCRIPTION:
Study to evaluate the bioequivalence of orally administered bosentan preparations, immediate release tablets, 125 mg in normal healthy subjects under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Healthy male aged 18 to 45 years.
* Verified diagnosis is "healthy" according to data Standard clinical, laboratory and Instrumental methods of examination.
* Have a body mass index between 18,5 and 30 kg/m2.
* Subjects must use, with their partner, methods of highly effective contraception throughout the study and 30 days after the end of study.
* Ability to keep fasting state for at least 14 hours.
* Consent and ability to respect the schedule of visits and the points of the Protocol.

Exclusion Criteria:

* History of serious allergic problems/events.
* Medicinal intolerance.
* Any acute and chronic diseases of the cardiovascular system, cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys, blood.
* Psychiatric disorders, history of epilepsy and seizures.
* Acute infectious diseases in less than 4 weeks before the start of the study.
* Subjects who have taken medication 2 weeks preceding before the study.
* Subjects who have taken any drugs known effects on hemodynamics or to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication (examples of inducers: barbiturates, omeprazole, etc.).
* Donation of plasma (450 mL or more) within 2 month prior to administration of the study medication.
* History of significant alcohol or drugs abuse or any indication of the regular use of more than 10 units of alcohol per week (1 Unit = 200 mL of wine or 500 mL of beer or 50 mL of alcohol 40%).
* Smokers.
* Participation in other clinical training is less than than for 3 months before the study.
* Lack of signed informed consent form.
* 10% deviation from references in lab tests.
* Positive testing for alcohol, drugs.
* Dehydration due to diarrhea, vomiting, or other causes within the last 24 hours before the start of the study.
* Any diet (vegetarian, etc.) extreme physical exercise, night shift work.
* Heart rate below 60 or above 80 beats per minute.
* Systolic blood pressure less than 110 mm Hg or more than 139 mm Hg.
* Diastolic blood pressure less than 60 mm Hg or more than 89 mm Hg.
* Volunteers, for Investigator opinion, who can not understand and evaluate the information about this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hours (pre-dose), as well as at 0.5, 1, 1.5, 2, 2.5, 3, 3,5, 3,75, 4, 4.25, 4.5, 4.75, 5, 6, 8, 10, 12, 14 and 24 hour post-dose.
  Pharmacokinetics of bosentan by Assessment of Observed Maximum Plasma Concentration (Cmax)
AUC(0-t) | 0 hours (pre-dose), as well as at 0.5, 1, 1.5, 2, 2.5, 3, 3,5, 3,75, 4, 4.25, 4.5, 4.75, 5, 6, 8, 10, 12, 14 and 24 hour post-dose.
  Pharmacokinetics of bosentan by Assessment of Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t))

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital № 3, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No